CLINICAL TRIAL: NCT02423005
Title: A Single-blind, Multi-centre, Randomised, Controlled, Non-inferiority, Clinical Study to Assess the Safety and Performance of the Neurotech Vital Compact Device Compared to the Itouch Sure Pelvic Floor Exerciser for the Treatment of Stress Urinary Incontinence in Female Patients
Brief Title: Neurotech Vital Compact Versus Itouch Sure Pelvic Floor Exerciser US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Therapeutics (Other)
Collaborators: Bio-Medical Research, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMR-13-1001
Record Dates: First submitted 2015-04-17; First posted 2015-04-22 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress urinary incontinence; Neurotech Vital Compact; 1h Provacative Pad Test; Neuroelectrical Muscle Stimulation (NEMS)
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Neurotech Vital Compact (Experimental): The Neurotech Vital Compact will be used by subjects with Stress Urinary Incontinence 5 days per week for 30 minutes per session for 12 weeks followed by 14 weeks of Kegel exercises.
  Interventions: Device: Neurotech Vital Compact
- itouch Sure Pelvic Floor Exerciser (Active Comparator): The itouch Sure Pelvic Floor Exerciser will be used by subjects with Stress Urinary Incontinence 7 days per week for 20 minutes per session for 12 weeks followed by 14 weeks of Kegel exercises.
  Interventions: Device: itouch Sure Pelvic Floor Exerciser

INTERVENTIONS:
Device: Neurotech Vital Compact — Neuromuscular electrical stimulation of the pelvic floor via an arrangement of external electrodes held in place by a garment.
  Arms: Neurotech Vital Compact
Device: itouch Sure Pelvic Floor Exerciser — Vaginal probe with electrodes designed to deliver electrical stimulation to the pelvic floor muscles.
  Other Names: EmbaGYN
  Arms: itouch Sure Pelvic Floor Exerciser

SUMMARY:
A prospective, randomised, controlled, single-blind, multi-site clinical study employing Neuromuscular Electrical Stimulation (NMES) to stimulate the pelvic floor muscles of women suffering from stress urinary incontinence.

Approximately one-hundred and eighty (180) female patients diagnosed with stress urinary incontinence will be enrolled in this study. All patients who are considered eligible to participate in the clinical study and give consent will be randomised to complete either a 12-week treatment programme with the Neurotech Vital Compact device or a 12-week treatment programme with the itouch Sure Pelvic Floor Exerciser. The 12-week treatment programme will be completed by the subjects at home with treatment with the device in accordance with the device Instructions for Use.

DETAILED DESCRIPTION:
This is a prospective, randomised, controlled, single-blind, multi-site clinical study to be conducted in the United States of America (USA) employing Neuromuscular Electrical Stimulation (NMES) to stimulate the pelvic floor muscles of women suffering from stress urinary incontinence.

Approximately one-hundred and eighty (180) female patients diagnosed with stress urinary incontinence will be enrolled in this study. All patients who are considered eligible to participate in the clinical study and give consent will be randomised to complete either a 12-week treatment programme with the Neurotech Vital Compact device or a 12-week treatment programme with the itouch Sure Pelvic Floor Exerciser. The 12-week treatment programme will be completed by the subjects at home with treatment with the device in accordance with the device Instructions for Use.

Subjects included in the clinical study will be evaluated at screening, on enrolment into the study (baseline) and during the 12-week treatment programme at 4 and 12 weeks. A telephone call will be made at 1 week to check on the patient's progress. In addition, subjects will be evaluated at 26 week following their commencement of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are female and at least 18 years of age, and not more than 65 years of age.
2. Subjects who have signed the informed consent form prior to any study related activity.
3. Subjects who have previously tried and failed to improve their condition using Kegel exercises.
4. Subjects who have been clinically diagnosed with stress urinary incontinence and demonstrate a greater than or equal to 3g urine leakage and a less than or equal to 90g urine leakage (>3g and < 90g) following a bladder-filling protocol and then a standardised stress test (provocative pad weight test) at the baseline assessment.
5. Subjects who score 9 or less (<9) out of 18 for the Urge Incontinence Questions and are confirmed as having predominant stress urinary incontinence on the Medical, Epidemiologic and Social Aspects of Aging Urinary Incontinence (MESA) Questionnaire completed at the screening assessment.
6. Subjects with a Body Mass Index of ≤ 35 kg/m2.
7. Subjects of child-bearing potential who are using a highly effective contraceptive method (established use of oral, injected, implanted hormonal method of contraception or barrier method of contraception with spermicide).
8. Subjects who are willing not to seek any other treatment for stress incontinence during the study period.
9. Subjects who are able to give voluntary, written informed consent to participate in this study and from whom consent has been obtained.
10. Subjects who are able to understand this study and are willing to complete all the study assessments.

Exclusion Criteria:

1. Subjects who have an existing medical condition that would compromise their participation in the study, e.g. reduced sensory perception in the contact area of the stimulation electrodes; scars or vaginal tissue wounds, lesions or inflamed/infected areas in the contact area of the stimulation electrodes; vaginal bleeding between menstrual periods; uncontrolled diabetes.
2. Subjects who have a physical condition that would make them unable to perform the study procedures, e.g. pelvic or hip surgery within the past 6 weeks.
3. Subjects who have been diagnosed with Chronic Obstructive Pulmonary Disease (COPD).
4. Subjects with a history of an underlying neurological condition, e.g. Multiple Sclerosis, Parkinson's disease, epilepsy.
5. Subjects with any bladder abnormality that would affect the urinary flow through the lower urinary tract including signs or symptoms of an active urinary tract infection, abnormal bladder capacity (e.g., >300 cc), post void residual volume >200 cc, spastic bladder, vesico-ureteral reflux or bladder stones.
6. Subjects with a blood clotting disorder or who are taking anti-coagulant medications.
7. Subjects who have previously had any uro-gynaecological related surgery that would affect the pelvic floor muscles or urinary flow through the urethra (excluding hysterectomy).
8. Subjects who have previously had pelvic floor radiation.
9. Subjects who have previously been treated for stress incontinence with injectable bulking agents and/or vaginal probes within the past 6 months.
10. Subjects with a clinical diagnosis of prolapse greater than Stage 2.
11. Subjects who are pregnant or could be pregnant.
12. Subjects who are less than 6 months post-partum or who are lactating.
13. Subjects who have any conductive intra-uterine devices or metal implants in the pelvic area, including hip and lumbar spine.
14. Subjects with pelvic pain or fibromyalgia or paravaginal defect.
15. Subjects with an active implanted medical device (i.e. pacemaker, insulin pump etc.) or conditions that may be adversely affected by electrical stimulation (e.g. cardiac arrhythmias).
16. Subjects with a current or active history of pelvic cancer and/or subjects with a life expectancy of less than 12 months.
17. Subjects who are currently involved in any injury litigation claims.
18. Subjects who have participated in a clinical study in the last 3 months or any previous clinical study with Bio-Medical Research Ltd.
19. Subjects who have been committed to an institution by virtue of an order issued either by the courts or by an authority.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who have achieved >50% improvement on the provocative pad weight test. | 12 weeks
  Subjects will complete an in-office 1 hour provocative pad test to determine volume of urine leaked during the test.

SECONDARY OUTCOMES:
Between group comparison of mean change in urine leakage in a provocative pad weight test | 12 Weeks
  Comparison of change on 1 hour pad test for Vital Compact vs. itouch Sure
Within group comparison of mean change in urine leakage in the 1 hour pad weight test | 12 weeks
  Comparison of change in urine leakage for each treatment arm
Between group comparison of the mean improvement in the Incontinence Quality of Life Questionnaire (I-QOL) score | 12 weeks
  Comparison of change in I-QOL score between groups
Between group comparison of the proportion of subjects achieving dryness | 12 weeks
  The treatment arms will be compared regarding the proportion of subjects who leak less than 1 g at the 12 week 1 hour pad test.
Between group comparison of mean change in the number of incontinence episodes per day. | 12 weeks
  Between group comparison of mean change in the number of incontinence episodes per day using a 7-day voiding diary.
Between group mean change in urine leakage in the 24-hour pad weight test | 12 weeks
  Between group comparison of mean change, with respect to baseline, in urine leakage in the 24-hour pad weight test
Within Neurotech Vital Compact group estimate of mean change in urine leakage in the 24-hour pad weight | 12 weeks
  • Within Neurotech Vital Compact group estimate of mean change, with respect to baseline, in urine leakage in the 24-hour pad weight
Within Neurotech Vital Compact group estimate of mean improvement in Incontinence Quality of Life Questionnaire (I-QOL) score | 12 weeks
  Within Neurotech Vital Compact group estimate of mean improvement, with respect to baseline, in Incontinence Quality of Life Questionnaire (I-QOL) score
Between group comparison of mean change in the number of pads used/day | 12 weeks
  Between group comparison of mean change, with respect to baseline, in the number of pads used/day recorded using a 7-day voiding diary
Within Neurotech Vital Compact group estimate of mean change in the number of pads used/day | 12 weeks
  Within Neurotech Vital Compact group estimate of mean change, with respect to baseline, in the number of pads used/day recorded using a 7-day voiding diary
Between group comparison of the proportion of subjects achieving dryness at Week 12 (<1g on the provocative pad weight test) | 12 weeks
  Between group comparison of the proportion of subjects achieving dryness at Week 12 (<1g on the provocative pad weight test)
Comparison of adverse events | 6 months
  Comparison between groups of adverse events reported throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Conor Minogue, PhD, Study Director — Bio-Medical Research, Ltd.
Locations (12):
- United States (12):
  - Maricopa Integrated Health Systems, Phoenix, Arizona
  - University of California Irvine Medical Center, Orange, California
  - Hartford Hospital, Hartford, Connecticut
  - Altus Research, Lake Worth, Florida
  - University of South Florida Medical Center, Tampa, Florida
  - Boston Clinical Trials, Boston, Massachusetts
  - AccuMed Research Associates, Garden City, New York
  - Lyndhurst Gynecological Associates, Winston-Salem, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The Jackson Clinic, Jackson, Tennessee
  - Renaissance Health & Surgical Associates, South Pittsburg, Tennessee

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2015-03-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT02423005/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2016-01-22): https://cdn.clinicaltrials.gov/large-docs/05/NCT02423005/SAP_001.pdf